CLINICAL TRIAL: NCT06813157
Title: Single-arm, Single-center Clinical Study of Mesenchymal Stem Cells in the Treatment of Refractory Primary Immune Thrombocytopenia
Brief Title: Mesenchymal Stem Cells in the Treatment of Refractory Primary Immune Thrombocytopenia
Acronym: MSC、ITP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-24-007; TXCE-2024-027 (Other: Dongguan Taixin Hospital Medical Ethics Committee)
Record Dates: First submitted 2025-01-19; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: ITP - Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: The subjects voluntarily signed the informed consent form, and after the evaluation of the screening period and the baseline period, they received 5 times of mesenchymal stem cell infusion in the treatment period, with a dose of 1 × 108/kg mesenchymal stem cells per time, with a frequency of 1 week between the first infusion and the second infusion (a time window of ±1 day), and the 3rd, 4th and 5th infusion were all 2 weeks apart from the last infusion (a time window of ±3 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSCs Injection (Experimental): The subjects voluntarily signed the informed consent form, and after the evaluation of the screening period and the baseline period, they received 5 times of mesenchymal stem cell infusion in the treatment period, with a dose of 1 × 108/kg mesenchymal stem cells per time, with a frequency of 1 week between the first infusion and the second infusion (a time window of ±1 day), and the 3rd, 4th and 5th infusion were all 2 weeks apart from the last infusion (a time window of ±3 days).
  Interventions: Other: MSC

INTERVENTIONS:
Other: MSC — The overall test process is as follows: screening period (V1): sign ICF, check the screening period, judge the criteria, record the baseline demographic information and the status of the subjects. Baseline period (V2): pre-transfusion assessment was performed to record the safety and other examinations of the subjects. During the treatment period (V3): according to the method and dose specified in the scheme, MSCs was treated for 5 times. Follow up period (V5): Safety and efficacy follow-up will be conducted at D14, M1, M2, M3, M6, M9, and M12 during the follow-up period.The subjects were followed up to M12 or those who met the withdrawal criteria withdrew early, whichever occurred first.

SUMMARY:
This study is a clinical study initiated by single-arm, single-center, multiple administration researchers. The main purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells in refractory ITP subjects. The subjects voluntarily signed the informed consent form, and after the evaluation of the screening period and the baseline period, they received 5 times of mesenchymal stem cell infusion in the treatment period, with a dose of 1 × 108/kg mesenchymal stem cells per time, with a frequency of 1 week between the first infusion and the second infusion (a time window of ±1 day), and the 3rd, 4th and 5th infusion were all 2 weeks apart from the last infusion (a time window of ±3 days). After all treatments were completed, the safety and effectiveness of D14, M1, M2, M3, M6, M9 and M12 were evaluated during the follow-up period. The subjects were followed up to M12 or those who met the withdrawal criteria withdrew early, whichever occurred first.

DETAILED DESCRIPTION:
The overall test process is as follows: screening period (V1): sign ICF, check the screening period, judge the criteria, record the baseline demographic information and the status of the subjects. Baseline period (V2): pre-transfusion assessment was performed to record the safety and other examinations of the subjects. During the treatment period (V3): according to the method and dose specified in the scheme, MSCs was treated for 5 times. Follow up period (V5): Safety and efficacy follow-up will be conducted at D14, M1, M2, M3, M6, M9, and M12 during the follow-up period.The subjects were followed up to M12 or those who met the withdrawal criteria withdrew early, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily signed the informed consent form;
2. The age is from 4 to 75 years old (including the critical value), male or female;
3. Patients clinically diagnosed as ITP (meeting the diagnostic criteria of the Chinese guidelines for the diagnosis and treatment of Primary immune Thrombocytopenia in Adults (2020 Edition)) had persistent thrombocytopenia for more than 3 months, but were ineffective to first-line drugs, second-line drugs for platelet production and rituximab, or ineffective to splenectomy / recurrence after operation.
4. Patients who received other maintenance regimens (including but not limited to corticosteroids, azathioprine, danazol or mycophenolate mofetil), but the stable dose had been maintained for at least 4 weeks, and the dose should remain unchanged during the trial period;
5. During screening, the liver and kidney function of the subjects met the following criteria: alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) ≤ 3 times of the upper limit of the normal value; total bilirubin ≤ 1.5 times of the upper limit of the normal value; creatinine ≤ 1.5 times of the upper limit of the normal value or creatinine clearance rate & gt; 75ml / min;
6. Women of childbearing age must have negative blood or urine pregnancy tests and are not breast-feeding, and agree to use medically approved contraceptive measures (such as intrauterine devices, condoms or contraceptive) during the study period.
7. Fertile male patients must agree to use barrier contraception or physical abstinence during the study;
8. The subjects were able to understand the nature and purpose of the trial, including possible risks and side effects, and to understand the researchers' oral and written medical orders and comply with the requirements of the trial.

Exclusion Criteria:

1. Have a history of severe allergic diseases or are allergic to research drugs;
2. There may be a history of angina pectoris, myocardial infarction, heart failure, severe arrhythmia, etc.
3. Combined use of anticoagulants or antiplatelet drugs;
4. In the first study, he was treated with gamma globulin within 2 weeks before medication.
5. The first study received rituximab within 24 weeks before treatment;
6. Other clinical trial drugs were used within 1 month before the use of drugs in the first study.
7. Uncontrolled hypertension (blood pressure is still higher than 160/100mmHg after active treatment);
8. Have a history of malignant tumor;
9. Those with a history of hepatitis B, or hepatitis C, or HIV, or immunodeficiency, or positive results of laboratory tests (hepatitis B surface antigen, or hepatitis C antibody, or HIV antibody) during screening;
10. Active / latent tuberculosis infection or other pathogen infection;
11. Live attenuated vaccine was vaccinated within 1 month before drug use in the first study, or there was a live attenuated vaccine program during the study period;
12. Hypogammaglobulinemia (IgG<400mg/dl) or IgA deficiency (IgA<10mg/dl);
13. History of important organ transplantation;
14. Patients with a history of severe mental illness;
15. The researchers believe that it is not appropriate for patients to participate in other conditions of this trial.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet count | From enrollment to the end of treatment at 12 moonths
  During the follow-up period, D14, M1, M2, M3, M6, M9, M12 were detected by blood routine test, and the changes of platelet count were observed.

SECONDARY OUTCOMES:
ITP Hemorrhage scale | From enrollment to the end of treatment at 12 months
  During the follow-up period, D14, M1, M2, M3, M6, M9, M12 were scored.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan Taixin Hospital, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial, only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code